CLINICAL TRIAL: NCT04415255
Title: Novel Use of Extrapleural Autologous Blood Injection in CT-guided Percutaneous Lung Biopsy and Its Comparison to Intraparenchymal Autologous Blood Patch Injection: A Single-center, Prospective, Randomized, and Controlled Clinical Trial
Brief Title: Novel Use of Extrapleural Autologous Blood Injection in CT-guided Percutaneous Lung Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Yasar Turk, Assistant Professor, Namik Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-AKD-150; 13.07.2018 1.0 (Other: Tekirdağ NKU Clinical Research Ethics Committee)
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Lung Biopsy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EPABI & IABPI (Experimental): extrapleural autologous blood injection (EPABI) along with intraparenchymal autologous blood patch injection (IABPI)
  Interventions: Other: EABPI plus IABPI
- IABPI-alone (Active Comparator): intraparenchymal autologous blood patch injection (IABPI)
  Interventions: Other: IABPI-alone

INTERVENTIONS:
Other: EABPI plus IABPI — If the patient was assigned to EPABI plus IABPI, while the extrapleural space was reached, ~ 15 ml of autologous blood was injected at the extrapleural space through the coaxial needle. Then the central stylet was reinserted and the coaxial needle was advanced into the lung parenchyma with a single puncture. The needle was stopped inside the proximal part of the target and the center needle was removed. A 20-G/16 cm fully-automated biopsy needle was introduced through the 19-G/13.8 cm coaxial needle and specimens were identically obtained. After specimens were collected, the biopsy needle was removed, and immediately the remaining autologous blood (~5 ml) was slowly injected through the coaxial needle as it was withdrawn through the parenchyma thus sealing the needle tract.
  Arms: EPABI & IABPI
Other: IABPI-alone — If the patient was assigned to IABPI-alone, after collecting the biopsy specimens, immediately the autologous blood (~5 ml) was slowly injected through the coaxial needle as it was withdrawn through the parenchyma thus sealing the needle tract.
  Arms: IABPI-alone

SUMMARY:
The purpose of this study is to evaluate the rate of iatrogenic pneumothorax and the need for intervention with extrapleural autologous blood injection (EPABI) along with intraparenchymal autologous blood patch injection (IABPI) or IABPI-alone in CT-guided percutaneous lung biopsy.

DETAILED DESCRIPTION:
The mechanism of pneumothorax is postulated to be due to the air leakage through the puncture hole when the needle is removed after the biopsy. However, pneumothorax may occur during the needle insertion as the visceral pleura is punctured or during the biopsy procedure before needle removal. Prevent such leakage, the investigators planned to inject autologous blood into the extrapleural space to prevent pneumothorax during needle entry. The extrapleural autologous blood injection (EPABI) is expected to form a space-occupying hematoma pressing on visceral pleura as a sealant. The investigators planned to test the EPABI method in a prospective single-center randomized controlled study design.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Referred for CT guided biopsy of lung lesion
* Target lesion of any size
* Target lesion located any away from visceral pleura based on the needle path
* Needle path without transgression of a pleural fissure, bleb, or bulla is possible
* Coaxial biopsy technique using Bard 19-Gauge introducer needle
* Needle length =16

Exclusion Criteria:

* Passage through non-aerated lung or tissue
* More than 1 biopsy on the same side requiring more than 1 pleural puncture
* History of prior ipsilateral lung interventions including:

Chest tube placement Surgery Pleurodesis Radiation treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the rate of iatrogenic pneumothorax and the need for intervention with extrapleural autologous blood injection (EPABI) | 1 years
  the rate of pneumothorax

CONTACTS AND LOCATIONS:
Overall Officials: Yasar Turk, Principal Investigator — Namik Kemal University
Locations (1):
- Tekirdag Namik Kemal University Medical Faculty Radiology Department, Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No